CLINICAL TRIAL: NCT05930912
Title: Psychiatric Orders in Psychoanalytic Treatment of ASD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yang I. Pachankis, PhD (Individual)
Collaborators: S for Science (Unknown)
Responsible Party: Sponsor-Investigator, Yang I. Pachankis, PhD, PI, Pachankis, Yang I., M.D.
Organization: Pachankis, Yang I., M.D. (Individual)
Other Study IDs: ASD-Psy-000; ASD-000000 (Other Grant/Funding Number: S for Science)
Record Dates: First submitted 2023-06-11; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: PTSD; Autism Spectrum Disorder High-Functioning; OCD; Agoraphobia With Panic Attacks; Depression, Unipolar; Depression, Anxiety; Depression and Suicide; Depression, Reactive; Depression; Psychoneurotic; Depression Anxiety Disorder; Panic Disorder With Agoraphobia, Severe Agoraphobic Avoidance and Mild Panic Attacks; Anxiety Disorders; ADHD - Combined Type; Borderline Personality Disorder; Social Anxiety Disorder; Avoidant Personality Disorder; Stockholm Syndrome; Grief; Separation Insecurity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder; Depression; Anxiety Disorders; Suicide; Adjustment Disorders; Borderline Personality Disorder; Phobia, Social; Personality Disorders | interventions — Sertraline; Duloxetine Hydrochloride; Serotonin and Noradrenaline Reuptake Inhibitors; Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participant Case: The participant started taking SNRI duloxetine 20 mg/night in Jan. 2023, and changed to SSRI sertraline 50 mg/d in Mar. 2023. The apparent positive psychedelic effects did not take effect until increased dosage to sertraline 100mg/d after around one week in Jun. 2023. Duloxetine is planned to be added to the mix thereon.
  Interventions: Diagnostic Test: Psychoanalysis; Drug: sertraline 50mg; Drug: Duloxetine 20 MG; Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Diagnostic Test: Psychoanalysis — Case-specific psychoanalysis is performed, including the participant's background during birth.
  Other Names: Psychodynamic analysis
Drug: sertraline 50mg — After the initial assessment of 50 mg/d, the treatment dosage is determined at 100 mg/d.
  Other Names: SSRI
Drug: Duloxetine 20 MG — Duloxetine is used with 20 mg/night for subsidiary effects with sertraline.
  Other Names: SNRI
Behavioral: Cognitive Behavioral Therapy — CBT is tailored to the participant's current activities and life decisions.
  Other Names: CBT

SUMMARY:
Autism Spectrum Disorder (ASD) is often accompanied by a variety of other symptoms, such as bipolar disorder, Attention Deficit Hyperactivity Disorder (ADHD), Social Anxiety Disorder (SAD), Avoidant Personality Disorder (AvPD), Obsessive Compulsive Disorder (OCD), etc. The behavioral and social complications often marginalize the population, impact on life satisfaction, undermined societal values that impact on economic and financial fairness, and so forth. Furthermore, persons with ASD are neurodiverse from standardized pharmacological and clinical cares, and are interpreted disadvantaged in the context of neurotypical treatments.

The research protocol aims to differentiate the neuropharmacological implications of ASD from its behavioral and social implications. Such a differentiation is beneficial to the quality of care for neurodiverse population, both in terms of precision treatment in medical settings, and in terms of psychotherapeutic treatment efficacy in the interpretation of behavioral and social traits.

The study protocol continues from the adverse event of the participant in NCT05711810 trial, after the positive immunological results in the NCT05839236 trial. The intervention medicine continues from Sertraline adjusted on the choice of Selective Serotonin Reuptake Inhibitor (SSRI) in the previous two trials for complex post-traumatic stress disorder (CPTSD) of the participant, and its combined used with Duloxetine in the choice of Selective Norephedrine Reuptake Inhibitor (SNRI) for norephedrine regulations.

The hypothesized target is on the discrete psychiatric intervention centered approach to ASD treatment care. In the PRC where the study is being carried out, amphetamine class medicines are strictly prohibited and defined as illegal substances, regardless of their only proven effect for ASD patient care. Contributed by the sociostructural elements and necessities, black market amphetamine and ketamine have not only emerged in the regime for decades, but also have become a lucrative business. Their recreational uses are also sometimes accompanied by real necessities and needs; black markets cater to the needs but guidance on the usages is based on word-of-mouth stories without professional medical assistances. There is one case the Principal Investigator (PI) collected, that one person, possibly under depression contributed by PTSD, took relatively high dosage of amphetamine and went into a state of psychosis with overwhelming persecution mania. The study protocol, Psychiatric Orders in Psychoanalytic Treatment of ASD, is therefore designed for an evidence-based approach in treating complex psychiatric disorders with psychoanalytic guidance.

ELIGIBILITY:
Inclusion Criteria:

* Persons with ASD.

Exclusion Criteria:

* Severe ASD cases with central nerve system complications.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is currently Asian, and the sociostructural environment of People's Republic of China is implied.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | 90 days
Generalized Anxiety Disorder (GAD-7) | 90 days
Dissociative Experiences Scale - II (DES-II) | 90 days
The Defeat Scale (D Scale) | 90 days
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 90 days
Severity Measure for Agoraphobia-Adult | 90 days
BPD Check List | 90 days
Rosenberg Self-Esteem Scale (RSE) | 90 days
Young Schema Questionnaire (YSQ) | 90 days
Personality Belief Questionnaire (PBQ) | 90 days
Behavioral Satisfaction Questionnaire (X axis) | 90 days
  The X axis score total range -150 to +140, from self-centrism (passive-aggressiveness) to proactive social behaviors.
Behavioral Satisfaction Questionnaire (Y axis) | 90 days
  The Y axis score total range -200 to +195, from inhibition to excitation of the hypothalamic-pituitary-adrenal (HPA) axis in daily lives.

SECONDARY OUTCOMES:
Heart Rate | 90 days
  Heart rate is used to correlate to the participant's mode change.
Systolic Blood Pressure | 90 days
  Systolic blood pressure is measured for reference on psychoneurotic correlations.
Diastolic Blood Pressure | 90 days
  Diastolic blood pressure is measured for reference on possible side-effects with dizziness etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Residential Address, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD is being shared on Open Science Framework with the DOI: 10.17605/OSF.IO/2MGJK.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available during the study process, and the archives after completion will stay available.
Access Criteria: Public.
URL: http://doi.org/10.17605/OSF.IO/2MGJK

REFERENCES:
- [Background] Yang IP. Questions of COVID-19: Institutional Derogations of Global Health. Lambert Academic Publishing. 2023. ISBN: 978-6206153849.
- [Background] Pachankis Y. Jeopardies in human security and politicization of COVID-19. Ethics Med Public Health. 2023 Apr;27:100871. doi: 10.1016/j.jemep.2023.100871. Epub 2023 Feb 1. No abstract available. PMID 36743192
- [Background] Yang IP. Dictatorial Psychopathological Commination in Server-Side Public Mental & Psychological Menace. Biomedical Science and Clinical Research. 2023; 2(2): 173-184.
- [Background] Yang IP. Proton Paths of Cardiac Immune Reflex. Online Journal of Cardiology Research & Reports. 2023; 7(1): 000655.
- [Background] Yang IP. What Do We Need in Adolescence?. Journal of Addiction Research. 2023; 7(1): 7-8.
- [Background] Yang IP. Proton Decay Reconstruction in Conscious Phenomenon - Literature Review on MRI, EEG, and PET Technologies. Advances in Sexual & Reproductive Health Research. 2022; 1(1): 128-130.
- [Background] Yang IP. Correlating Nuclear Sciences to Biochemistry - Mini-review on the Environmental Physiological Impact of Electronic Warfare on Public Health. Journal of Clinical Chemistry. 2022; 1(2): 1-5.
- [Background] Yang IP. Mass Surveillance, Behavioural Control, and Psychological Coercion - The Moral Ethical Risks in Commercial Devices. In: Wyld, D. C. & Nagamalai, D. (Eds.) Computer Science and Information Technology. 2022; 151-168. AIRCC Publishing Corporation.
- [Background] Yang IP. Technical Analysis on the Cyber Organizational Criminology of Dictatorial Military Conducts -- Experience from Human Trafficking and Coercions by Military Cyber Aggressions. International Journal of Security, Privacy and Trust Management. 2022; 11(3): 1-19.
- [Background] Yang IP. The Cultural Revisionist Element behind P. R. China's Neo-Nazism: A Cross-cultural and Cross-religion Research. International Journal of Advanced Multidisciplinary Research and Studies. 2022; 2(4): 435-451.
- [Background] Yang IP. A Self--help Guide to Psychoanalysis in Cisgender Homosexual Male. Journal of Marketing Management and Consumer Behavior. 2022; 4(2), 93-110.
- [Background] Yang IP. An Evidence-driven Research to the Transgressions of Geneva Conventions by the Communist Party of China Led Autocratic Regime. International Journal of Scientific & Engineering Research. 2022; 13(10): 249-266.
- [Background] Yang IP. Targeted Human Trafficking - The Wars between Proxy and Surrogated Economy. International Journal of Scientific & Engineering Research. 2022; 13(7): 398-409.
- [Background] Yang IP. Why Should LGBTQI Marriage Be Legalized. Academia Letters. 2022; Article 5157.
- Available data/document: Individual Participant Data Set — http://doi.org/10.17605/OSF.IO/2MGJK
- Available data/document: Social Circumstances and Events: zenodo.7382529 — http://doi.org/10.5281/zenodo.7382529
- Available data/document: Cyber-Social Circumstances and Events: zenodo.6942208 — http://doi.org/10.5281/zenodo.6942208
- Available data/document: Social Circumstances and Events: zenodo.7188211 — http://doi.org/10.5281/zenodo.7188211
- Available data/document: Cyber-Social Circumstances and Events: zenodo.6941906 — http://doi.org/10.5281/zenodo.6941906
- Available data/document: Cyber-Social Circumstances and Events: zenodo.6952516 — http://doi.org/10.5281/zenodo.6952516
- Available data/document: Analytic Code: zenodo.7022873 — http://doi.org/10.5281/zenodo.7022873 — The technological-psychoanalytic mass psychological observation and analysis schemes.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT05930912/Prot_SAP_ICF_000.pdf